CLINICAL TRIAL: NCT01721317
Title: Study PTG116878, a Dose-Optimization Study of Ezogabine/Retigabine Immediate Release Tablets Versus Placebo in the Adjunctive Treatment of Subjects With Partial-Onset Seizures
Brief Title: Dose-Optimization, Adjunctive Treatment Study of Ezogabine/Retigabine Immediate Release in Partial-onset Seizures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After reevaluation of the benefit: risk profile of ezogabine/retigabine, GSK does not believe the early adjunctive treatment study population is appropriate.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116878; 2012-003105-10 (EudraCT Number)
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Seizures
Keywords: Ezogabine/Retigabine; Adjunctive Treatment; Safety; Efficacy; Epilepsy; Tolerability; Immediate Release; GW582892; Dose-Optimization; Partial-Onset Seizures
MeSH Terms: conditions — Seizures; Epilepsy | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (16):
- Titration Phase: Ezogabine/Retigabine 300 mg (Experimental): Subjects receive Ezogabine/Retigabine 300 mg equally divided TID over Wk 1
  Interventions: Drug: Ezogabine/Retigabine IR
- Titration Phase: Placebo 300 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Titration Phase: Ezogabine/Retigabine 450 mg (Experimental): Subjects receive Ezogabine/Retigabine 450 mg equally divided TID over Wk 2
  Interventions: Drug: Ezogabine/Retigabine IR
- Titration Phase: Placebo 450 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Dose-Optimization Phase: Ezogabine/Retigabine 600 mg (Experimental): Subjects receive Ezogabine/Retigabine 600 mg equally divided (200 mg TID) over Wk 3 or until they achieve their optimal tolerated dose as assessed by the Investigator
  Interventions: Drug: Ezogabine/Retigabine IR
- Dose-Optimization Phase: Placebo 600 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Dose-Optimization Phase: Ezogabine/Retigabine 750 mg (Experimental): Subjects receive Ezogabine/Retigabine 750 mg equally or unequally divided TID over Wk 4 or until they achieve their optimal tolerated dose as assessed by the Investigator
  Interventions: Drug: Ezogabine/Retigabine IR
- Dose-Optimization Phase: Placebo 750 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Dose-Optimization Phase: Ezogabine/Retigabine 900 mg (Experimental): Subjects receive Ezogabine/Retigabine 900 mg equally or unequally divided TID over Wk 5 or until they achieve their optimal tolerated dose as assessed by the Investigator
  Interventions: Drug: Ezogabine/Retigabine IR
- Dose-Optimization Phase: Placebo 900 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Dose-Optimization Phase: Ezogabine/Retigabine 1050 mg (Experimental): Subjects receive Ezogabine/Retigabine 1050 mg equally or unequally divided TID over Wk 6 or until they achieve their optimal tolerated dose as assessed by the Investigator
  Interventions: Drug: Ezogabine/Retigabine IR
- Dose-Optimization Phase: Placebo 1050 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Dose-Optimization Phase: Ezogabine/Retigabine 1200 mg (Experimental): Subjects receive Ezogabine/Retigabine 1200 mg equally divided (400 mg TID) over Wk 7 or until they achieve their optimal tolerated dose as assessed by the Investigator
  Interventions: Drug: Ezogabine/Retigabine IR
- Dose-Optimization Phase: Placebo 1200 mg (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo
- Maintenance Phase:Ezogabine/Retigabine (Experimental): Subjects receive Ezogabine/Retigabine at the daily dose achieved (equally or unequally divided TID) at the end of the Dose-Optimization Phase for 8 Weeks (600 mg, 750 mg, 900 mg, 1050 mg, or 1200 mg)
  Interventions: Drug: Ezogabine/Retigabine IR
- Maintenance Phase: Placebo (Placebo Comparator): Subjects receive matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezogabine/Retigabine IR — Subjects received drug (dose strength 300 mg to 1200 mg) orally with or without food. The 3 daily doses are to be administered with approximately an 8-hour interval between them.
  Arms: Dose-Optimization Phase: Ezogabine/Retigabine 1050 mg; Dose-Optimization Phase: Ezogabine/Retigabine 1200 mg; Dose-Optimization Phase: Ezogabine/Retigabine 600 mg; Dose-Optimization Phase: Ezogabine/Retigabine 750 mg; Dose-Optimization Phase: Ezogabine/Retigabine 900 mg; Maintenance Phase:Ezogabine/Retigabine; Titration Phase: Ezogabine/Retigabine 300 mg; Titration Phase: Ezogabine/Retigabine 450 mg
Drug: Placebo — Matching placebo will be available
  Arms: Dose-Optimization Phase: Placebo 1050 mg; Dose-Optimization Phase: Placebo 1200 mg; Dose-Optimization Phase: Placebo 600 mg; Dose-Optimization Phase: Placebo 750 mg; Dose-Optimization Phase: Placebo 900 mg; Maintenance Phase: Placebo; Titration Phase: Placebo 300 mg; Titration Phase: Placebo 450 mg

SUMMARY:
This is a Phase IV adjunctive treatment dose-optimization study evaluating the efficacy, safety, and health outcomes of ezogabine/retigabine immediate release (IR) (GW582892) compared with placebo in adult subjects with partial-onset seizures (POS). This randomized, double-blind, placebo-controlled, parallel-group, multicenter study will compare ezogabine/retigabine IR (investigator-selected daily doses of 600 milligram (mg)/day, 750 mg/day, 900 mg/day, 1050 mg/day or 1200 mg/day) with placebo. Study drug will be taken three times a day (TID) in equally or unequally divided doses.

The study design includes up to a 10-week (wk) Screening (≤2 wks)/Baseline (8 wks) Phase, a Titration Phase (2 wks), Dose-Optimization Phase (8 wks), Maintenance Phase (8 wks), and Taper/Follow-Up Phase (3 wks). The total duration of the study for each subject will be approximately 31 wks, and at minimum approximately 27 wks if subjects provide reliable 28-day retrospective seizure data.

Approximately 280 subjects will be screened with approximately 208 subjects randomly assigned to 1 of 2 treatment groups in a 2:1 ratio (ezogabine/retigabine IR, or placebo).

Subjects will be instructed to start investigational product (IP) the day after the baseline visit. During the first week of the Titration Phase, subjects will be taking 300 mg/day (100 mg TID). During the second week, subjects will be taking 450 mg/day (150 mg/day TID).

At the beginning of the Dose-Optimization Phase (3rd week of study drug) subjects will take 600 mg/day (200 mg TID) for one week. Thereafter during the Dose-Optimization Phase, subjects will continue to increase their daily dose by 150 mg per week until they have achieved their optimal tolerated dose. During this phase, the investigator may choose to have the subject stay on his/her designated dose for another week before attempting a dose increase until reaching a dose of 1200 mg/day. In addition, in the context of tolerability issues, the subject may be reduced to the preceding dose level for one week before attempting to increase the dose again at the next scheduled time point until the subject reaches optimal dose. Subjects unable to tolerate a minimum of 600 mg/day will be discontinued from the study.

The Maintenance Phase will begin at Week 10 (Visit 8) and will last 8 weeks. During the Maintenance Phase, subjects will remain on the daily TID dose achieved at the end of the Dose-Optimization Phase.

Seizure type and frequency will be monitored throughout the study via a Seizure Calendar and will be evaluated at each study visit. Subjects will be instructed to complete the daily Seizure Calendar during each phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* A male or female of 18 years of age or above capable of giving written informed consent
* Have a confident diagnosis of epilepsy for >=6 months with partial-onset seizures (POS), i.e., simple or complex POS with or without secondary generalization (classified according to the International League Against Epilepsy (ILAE) Guidelines, prior to the Screening Visit
* Currently receiving monotherapy treatment with an antiepileptic drug (AED) at a stable dose for at least 28 days prior to the screening visit (Visit 1). If the subject is taking a barbiturate (e.g., phenobarbital), the dose must be stable for ≥3 months prior to the Screening Visit. Note: Subjects who have received previous adjunctive treatment but are currently taking one AED are eligible for enrolment.
* Investigator-confirmed partial seizure frequency rate of ≥3 partial seizures per 28 days over the 8 weeks preceding the screening visit and must not have been seizure-free for ≥ 21 consecutive days.
* Female of non-child bearing potential, or female of child-bearing potential willing to use protocol-specified methods of contraception to prevent pregnancy during the study.
* Capable to comply with dosing of study drug, background AED, all study procedures and to maintain an accurate and complete daily written Seizure Calendar and Functional Status Diary

Exclusion Criteria:

* Have generalized epilepsy (e.g. Lennox-Gastaut, Juvenile Myoclonic epilepsy, Absence, etc.) or non-epileptic seizures.
* Have had innumerable seizures within the 12-month period prior to the Screening Visit where the individual seizures cannot be counted.
* Have had status epilepticus within 12 months prior to screening
* Have a history of pseudo seizures, non-epileptic events or any other type of psychogenic seizures that could be confused with seizures.
* Have been treated with felbamate or vigabatrin within the 6 months prior to Screening. If a subject has been previously treated with vigabatrin >6 months prior to Screening, a visual perimetry test performed within 6 months prior to Screening must show normal visual fields or no worsening of recognized visual field abnormalities as compared with prior to vigabatrin treatment
* Benzodiazepines used in any manner other than acute usage as defined in this protocol will be considered concurrent AED usage and will not be permitted

  * Are using Central Nervous System (CNS)-active medication (other than concomitant AED therapy), unless the subject has been stabilized on such medication for at least 1 month prior to the Screening Visit.
* Are using herbal treatments with CNS activity within at least 1 month prior to the Screening Visit
* Have received ezogabine/retigabine in a previous study or have taken POTIGA or TROBALT.
* Are currently following or planning to follow the ketogenic diet
* Have an active Vagus Nerve Stimulator (VNS) to control seizures
* Are planning surgery to control seizures during the study
* Have impaired renal function as judged by a creatinine clearance of <50 mL/min
* Have a history of urinary retention or risk factors for urinary retention that in the investigator's judgment could potentially affect subject safety.
* Have an average corrected QT interval (QTc), using Bazett's QT correction (QTcB), ≥450msec or ≥480msec for subjects with bundle branch block at the time of the Screening Visit
* Liver function tests: alanine aminotransferase (ALT) is ≥2 times the upper limit of normal (ULN); alkaline phosphatase and bilirubin are >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Are suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormalities that are likely to interfere with the objectives of the study
* Have a history of malignancy within the past 2 years; with the exception of basal cell carcinoma
* Have unstable liver disease [chronic stable hepatitis B and C are acceptable if subject otherwise meets entry criteria; chronic stable Hepatitis B to be excluded if significant immunosuppressive agents administered due to risk of hepatitis B reactivation]
* Have any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect subject safety or study outcome, including but not limited to: clinically significant cardiac, renal, hepatic condition, or a condition that affects the absorption, distribution, metabolism or excretion of drugs
* Have an active suicidal plan/intent or have had active suicidal thoughts in the past 6 months. Have history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Have a history of substance abuse (alcohol or drugs) or substance dependence within 12 months prior to screening
* Have a known hypersensitivity to any components of the study medication
* Have taken an investigational drug, or used an investigational device, within the previous 30 days prior to screening or plans to take an investigational drug anytime during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2013-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (9):
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Golden Valley, Minnesota
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Kingwood, Texas
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, parallel-group, multicenter study comparing ezogabine/retigabine immediate release (IR) with placebo, as adjunctive treatment in adults with partial-onset seizures. The study was prematurely discontinued after randomizing only 6 of the planned 208 participants.
Pre-assignment Details: The study consisted of a 2-week (or less) Screening Phase, an 8-week Baseline Phase, a 2-week Titration Phase, an 8-week Dose-Optimization Phase, an 8-week Maintenance Phase, and a 3-week Taper Phase.
Groups:
- Placebo: Participants received matching ezogabine/retigabine IR placebo orally three times a day (TID) in equally or unequally divided doses.
- Ezogabine/Retigabine IR: Participants received investigator-selected daily doses of 600 milligrams (mg)/day, 750 mg/day, 900 mg/day, 1050 mg/day or 1200 mg/day of ezogabine/retigabine IR. The study drug was taken orally TID in equally or unequally divided doses.
Period: Overall Study
Arm/Group | Placebo | Ezogabine/Retigabine IR
Started | 2 | 4
Completed | 0 | 0
Not Completed | 2 | 4
Not completed — Study Closed / Terminated | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching ezogabine/retigabine IR placebo orally TID in equally or unequally divided doses.
- Ezogabine/Retigabine IR: Participants received investigator-selected daily doses of 600 mg/day, 750 mg/day, 900 mg/day, 1050 mg/day or 1200 mg/day of ezogabine/retigabine IR. The study drug was taken orally TID in equally or unequally divided doses.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ezogabine/Retigabine IR | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (10.61) | 42.8 (16.32) | 42.7 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 28-day Total Partial Seizure Frequency (POS) From Week 0 (End of Baseline Phase) Through Week 18 (End of Maintenance Phase)
Description: The efficacy of ezogabine/retigabine IR as an adjunctive treatment was to be evaluated by the percent change in the total partial seizure frequency, which was recorded by participants in the daily seizure calendar. The total 28-day POS rate is defined as the total number of POS reported during the evaluation period divided by the total number of applicable days during the evaluation period with this quotient multiplied by 28 days. The applicable days are the days in which the participant had non-missing seizure data (i.e., either 0 or > 0 seizures recorded). Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase) through Week 18 (end of Maintenance Phase)
Population: Intent-to-Treat (ITT) Population: all randomized participants who received >= 1 dose of study medication and who had >= 1 post-Baseline seizure diary day with >= 0 seizures recorded.
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percent Change in the 28-day Total Partial Seizure Frequency (POS) Within Each Stratum From Week 0 (End of Baseline Phase) Through Week 18 (End of Maintenance Phase)
Description: The percent change in 28-day total POS frequency within each stratum (sodium channel blocker or non-sodium channel blocker) background antiepileptic drug (AED) was to be summarized as the supportive analysis. The total 28-day POS value is defined as the total number of POS reported during the evaluation period divided by the total number of applicable days during the evaluation period with this quotient multiplied by 28 days. The applicable days are the days in which the participant had non-missing seizure data (i.e., either 0 or > 0 seizures recorded). Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase) through Week 18 (end of Maintenance Phase)
Population: ITT Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change in 28-day Total Partial Seizure Frequency (POS) for the Indicated Intervals: Maintenance Phase and the Dose-Optimization Phase + Maintenance Phase
Description: The efficacy of ezogabine/retigabine IR as an adjunctive treatment was to be evaluated by the percent change in total partial seizure frequency during the Dose-Optimization Phase and Maintenance Phase. The total 28-day POS value is defined as the total number of POS reported during the evaluation period divided by the total number of applicable days during the evaluation period with this quotient multiplied by 28 days. The applicable days are the days in which the participant had non-missing seizure data (i.e., either 0 or > 0 seizures recorded). Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 3 (start of Dose -Optimization Phase) to Week 18 (end of Maintenance Phase)
Population: ITT Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Par. Experiencing >=50% Reduction in 28-day Total Partial Seizure Frequency (POS) for the Intervals: Double-blind Period (Titration Phase + Dose-Optimization Phase + Maintenance Phase), Maintenance Phase and Dose-Optimization + Maintenance Phase
Description: Participants (par.) experiencing >= 50% reduction from Baseline to the end of the Double-Blind Phase in 28-day total POS were to be reported. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase) through Week 18 (end of Maintenance Phase)
Population: ITT Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Seizure Free Participants for the Indicated Intervals: Maintenance Phase and the Dose-Optimization Phase + Maintenance Phase
Description: Participants without seizures during the interval of Maintenance Phase and the Dose-Optimization Phase + Maintenance Phase were to be reported. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 3 (start of Dose-Optimization Phase) to Week 18 (end of Maintenance Phase)
Population: ITT Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in the Number of Seizure Free Days for the Indicated Intervals: Double-blind Period (Titration Phase + Dose-Optimization Phase + Maintenance Phase), Maintenance Phase and the Dose-Optimization + Maintenance Phase
Description: The change in number of seizure free days during the Double-Blind period, the Maintenance Phase and the Dose-Optimization Phase + Maintenance Phase were to be reported. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase) to Week 18 (end of Maintenance Phase)
Population: ITT Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in Functional Status (Epilepsy-related Worry and Activity Limitation) and Productivity (Missed Work or School) to the End of the Dose-Optimization Phase and the End of the Maintenance Phase
Description: The effect of ezogabine/retigabine IR as an adjunctive treatment on health outcomes was to be evaluated on the basis of functional status and productivity. Participants were asked to complete the paper functional status diary to collect information to assess how the participant's functional status is affected by their epilepsy symptoms. Participants were asked to rate their epilepsy-related worry, activity limitations, and productivity (missed work or school). Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 3 (start of Dose -Optimization Phase) to Week 18 (end of Maintenance Phase)
Population: ITT Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Incidence of New Seizure Types in Participants Without a History of These Seizure Types
Description: The safety and tolerability of ezogabine/retigabine IR was to be evaluated by recording the incidence of new seizure types in participants without a history of these seizure types. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase) to Week 21 (end of Taper Phase)
Population: Safety Population: all randomized participants who receive >= 1 dose of study medication.
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants at Each Dose During the Maintenance Phase and Average Maintenance Dose Over All Participants
Description: The safety and tolerability of ezogabine/retigabine IR was to be evaluated by recording the number of participants at each dose during the Maintenance Phase and the average maintenance dose over all participants. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 11 (start of Maintenance Phase) to Week 18 (end of Maintenance Phase)
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Early Study Discontinuation
Description: The safety and tolerability of ezogabine/retigabine IR was to be evaluated by recording the incidence of participants with early study discontinuation.
Time Frame: Week 0 (end of Baseline Phase) to Week 21 (end of Taper Phase)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 2 | 4
Participants | 2 | 4

11. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from Baseline in body weight was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Screening, Week 0 (end of Baseline Phase), Week 2 (end of Titration Phase), Week 10 (end of Dose-Optimization Phase), Week 18 (end of Maintenance Phase) and Week 21 (end of Taper Phase)
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from Baseline in blood pressure was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 11
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Heart Rate
Description: Change from Baseline in heart rate was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 11
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in the QT Interval Using Bazett's Correction (QTcB) and QT Interval Using Fridericia's Correction (QTcF)
Description: Change from Baseline in the QT interval using Bazett's correction (QTcB) and QT interval using Fridericia's correction were to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 11
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in the Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Segmented Neutrophils and Red Blood Cell (RBC) Distribution Width
Description: The change from Baseline in the indicated hematology tests were to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Screening, Week 0 (end of Baseline Phase), Week 10 (end of Dose-Optimization Phase), Week 18 (end of Maintenance Phase) and Week 21 (end of Taper Phase)
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in the Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Segmented Neutrophils, White Blood Cell (WBC) Count and Platelet Count
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change From Baseline in Hematocrit
Description: The change from Baseline in the indicated hematology test was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count
Description: as for outcome 18
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin
Description: as for outcome 18
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change From Baseline in Albumin and Total Protein
Description: The change from Baseline in the indicated chemistry tests were to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase, Lactate Dehydrogenase and Gamma Glutamyltransferase (GGT)
Description: as for outcome 21
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Uric Acid and Creatinine
Description: as for outcome 21
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Change From Baseline in Calcium, Chloride, Potassium, Sodium, Glucose, Magnesium, Phosphorus Inorganic, Bicarbonate and Urea/Blood Urea Nitrogen (BUN)
Description: as for outcome 21
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Change From Baseline in BUN/Creatinine Ratio
Description: The change from Baseline in the indicated chemistry tests was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Change From Baseline in Creatinine Clearance
Description: The change from Baseline in the indicated chemistry test was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change From Baseline in Urine Specific Gravity (USG)
Description: The change from Baseline in the indicated urinalysis test was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: The change from Baseline in the indicated urinalysis test was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize ot evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Number of Participants for the Indicated Urinalysis Parameters Tested by Dipstick
Description: The change from Baseline in the following urinalysis parameters (urine occult blood, urine glucose, urine ketones and urine protein) were to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: as for outcome 15
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Change From Baseline in Post-void Residual (PVR) Urinary Bladder Ultrasound Volume
Description: The change from Baseline in the PVR bladder ultrasound results was to be assessed. Due to the study being prematurely terminated, there was not sufficient data to summarize or evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase), Week 10 (end of Dose-Optimization Phase) and Week 18 (end of Maintenance Phase)
Population: Safety Population
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Number of Participants With the Indicated Assessment Events of Suicidal Behavior, Suicidal Ideation or Non-suicidal Self Injurious Behavior Via the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Prospective assessment of suicidality was conducted using the Columbia-Suicide Severity Rating Scale (C-SSRS), a brief questionnaire designed to assess severity and change in suicidality by integrating both behavior and ideation using a semi-structured interview to probe participant responses. C-SSRS data were only collected through Week 8 for the 6 randomized participants. Due to the study being prematurely terminated, there was not sufficient data to evaluate this endpoint.
Time Frame: Week 0 (end of Baseline Phase), Week 2 (end of Titration Phase), Week 4, Week 6 and Week 8
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Ezogabine/Retigabine IR
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the investigational product until the Follow-up period (up to Study Day 147).
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | Ezogabine/Retigabine IR
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | Ezogabine/Retigabine IR (N=4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.